CLINICAL TRIAL: NCT05396963
Title: Effects of Egg White Supplementation on Body Composition, Physical Performance, and Amino Acid Profile of Individuals Undergoing High-intensity Functional Training
Brief Title: Egg White Supplementation in High-Intensity Functional Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: European Commission (Other); Greek Ministry of Development (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: EGGPROScience1
Record Dates: First submitted 2022-04-26; First posted 2022-05-31 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Exercise Training; Dietary Supplements
MeSH Terms: interventions — Egg White; Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are instructed not to disclose the supplement they are taking to their trainers, investigator, or outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Egg white - Whey protein - Maltodextrin (Other): Participants will receive egg white, whey protein, and maltodextrin in this order.
  Interventions: Dietary Supplement: Egg white; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Egg white - Maltodextrin - Whey protein (Other): Participants will receive egg white, maltodextrin, and whey protein in this order.
  Interventions: Dietary Supplement: Egg white; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Whey protein - Egg white - Maltodextrin (Other): Participants will receive whey protein, egg white, and maltodextrin in this order.
  Interventions: Dietary Supplement: Egg white; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Whey protein - Maltodextrin - Egg white (Other): Participants will receive whey protein, maltodextrin, and egg white in this order.
  Interventions: Dietary Supplement: Egg white; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Maltodextrin - Egg white - Whey protein (Other): Participants will receive maltodextrin, egg white, and whey protein in this order.
  Interventions: Dietary Supplement: Egg white; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Maltodextrin - Whey protein - Egg white (Other): Participants will receive maltodextrin, whey protein, and egg white in this order.
  Interventions: Dietary Supplement: Egg white; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Egg white — Intake of egg white
Dietary Supplement: Whey protein — Intake of whey protein
Dietary Supplement: Maltodextrin — Intake of maltodextrin

SUMMARY:
High-intensity functional training (HIFT), a new version of high-intensity interval training, has gained interest in recent years. HIFT is based on the CrossFit training template and includes multijoint movement patterns via both endurance and strengthening exercises. Research has shown positive effects of HIFT on body composition, cardiorespiratory fitness, and muscle performance of young individuals. The effectiveness of HIFT in higher ages and its protein requirements are less well documented. Protein requirements have been widely investigated in resistance training, where it has been found that protein supplementation may have additive beneficial effects on muscle strength and lean body mass. However, there is a research gap regarding the adaptations to HIFT when combined with protein supplementation.

Thus, the aim of this research is to compare the effects of egg white supplementation, whey protein supplementation (as a positive comparator), and maltodextrin (a carbohydrate as placebo) on body composition, physical performance, and plasma amino acid profile in young and middle-aged trained individuals of both sexes who perform HIFT. Participants will take all three supplements for 6 weeks each, with 2 weeks of washout (no supplementation) in between, in random and counterbalanced order. Researchers will not know the supplementation status of the participants. Participants will receive 0.6 g of protein or placebo per kg body weight daily on top of isoenergetic dietary plans to avoid differences in energy intake that might compromise the validity of the study. The dietary plans will be individualized and will provided 1.0 g protein/kg body weight/day. The HIFT protocol will include multimodal patterns of movement, combining endurance and strengthening exercises with the use of equipment such as Total Resistance eXercise (TRX), Bosu, kettlebells, and barbells.

Participants will undergo measurements of muscle strength, muscle endurance, aerobic capacity, and body composition at the beginning and end of the study, as well as during the two washout periods. Also, plasma amino acids, hematology, biochemistry, and hormones will be measured. Comparison of all these outcome measures between supplements will reveal whether protein supplementation is useful in HIFT.

ELIGIBILITY:
Inclusion Criteria:

* Regular training (mixed endurance and resistance training 3 to 6 times a week, 50 min each session, for the past 4 months), as assessed by gym records or questionnaires
* Clearance from a pathologist or cardiologist to perform maximal exercise
* Mixed isoenergetic diet for the past 4 months

Exclusion Criteria:

* Smoking (even one cigarette or nicotine-containing device over the past 6 months)
* Any injuries to the musculoskeletal system that could interfere with the execution of training
* Chronic disease
* Egg allergy
* Milk allergy
* Pregnancy, lactation, or planning a pregnancy within the duration of the study
* Regular use of prescription medicine or supplements that might affect muscle function or recovery over the past month
* Intermittent or religious fasting
* Any vegetarian, ketogenic or protein diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Lean and fat mass pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Lean and fat mass of the whole body and its parts (trunk, legs and arms) will be assessed by dual X-ray absorptiometry.
Lean and fat mass post-supplementation | Within 2 weeks after the end of supplementation.
  Lean and fat mass of the whole body and its parts (trunk, legs and arms) will be assessed by dual X-ray absorptiometry.
Maximal dynamic strength of shoulder muscles pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Maximal dynamic strength of shoulder muscles will be assessed by measurement of one-repetition maximum.
Maximal dynamic strength of shoulder muscles post-supplementation | Within 2 weeks after the end of supplementation.
  Maximal dynamic strength of shoulder muscles will be assessed by measurement of one-repetition maximum.
Force-velocity relationship of knee flexors and extensors pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Force-velocity relationship of knee flexors and extensors will be assessed in isokinetic dynamometer.
Force-velocity relationship of knee flexors and extensors post-supplementation | Within 2 weeks after the end of supplementation.
  Force-velocity relationship of knee flexors and extensors will be assessed in isokinetic dynamometer.
Plasma amino acid profile pre-supplementation | Within 4 days before the beginning of supplementation.
  Plasma amino acid profile (that is, the concentration of each individual amino acid) will be determined by liquid chromatography - mass spectrometry.
Plasma amino acid profile post-supplementation | Within 4 days after the end of supplementation.
  Plasma amino acid profile (that is, the concentration of each individual amino acid) will be determined by liquid chromatography - mass spectrometry.
Aerobic fitness pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Aerobic fitness will be assessed by measurement of maximal oxygen uptake through a maximal graded exercise test on treadmill.
Aerobic fitness post-supplementation | Within 2 weeks after the end of supplementation.
  Aerobic fitness will be assessed by measurement of maximal oxygen uptake through a maximal graded exercise test on treadmill.
Muscle endurance pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Muscle endurance will be assessed by performing multiple sit-ups, knee flexions and knee extensions.
Muscle endurance post-supplementation | Within 2 weeks after the end of supplementation.
  Muscle endurance will be assessed by performing multiple sit-ups, knee flexions and knee extensions.

SECONDARY OUTCOMES:
Biochemical analyses pre-supplementation | Within 4 days before the beginning of supplementation.
  Plasma glucose, triacylglycerols, total cholesterol, HDL cholesterol, LDL cholesterol, urea, and creatinine (all in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Biochemical analyses post-supplementation | Within 4 days after the end of supplementation.
  Plasma glucose, triacylglycerols, total cholesterol, HDL cholesterol, LDL cholesterol, urea, and creatinine (all in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Hormonal analyses pre-supplementation | Within 4 days before the end of supplementation.
  Plasma cortisol and testosterone (both in μg/dL) will be measured by immunoluminescence in an automated analyzer.
Hormonal analyses post-supplementation | Within 4 days after the end of supplementation.
  Plasma cortisol and testosterone (both in μg/dL) will be measured by immunoluminescence in an automated analyzer.
Resting metabolic rate pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Resting metabolic rate will be assessed with indirect calorimetry through the measurement of oxygen consumption with a metabolic analyzer.
Resting metabolic rate post-supplementation | Within 2 weeks after the end of supplementation.
  Resting metabolic rate will be assessed with indirect calorimetry through the measurement of oxygen consumption with a metabolic analyzer.
Internal load of exercise pre-supplementation | Within the first week of supplementation.
  Internal load of exercise will be assessed by telemetric heart rate sensors and software
Internal load of exercise post-supplementation | Within the last week of supplementation (week 6).
  Internal load of exercise will be assessed by telemetric heart rate sensors and software
Full blood count pre-supplementation | Within 4 days before the beginning of supplementation
  Full blood count will be performed by flow cytometry
Full blood count post-supplementation | Within 4 days after the end of supplementation.
  Full blood count will be performed by flow cytometry
Plasma enzymes pre-supplementation | Within 4 days before the beginning of supplementation.
  Creatine kinase and γ-glutamyltransferase (both in U/L) will be measured by chemiluminescence in an automated analyzer
Plasma enzymes post-supplementation | Within 4 days after the end of supplementation.
  Creatine kinase and γ-glutamyltransferase (both in U/L) will be measured by chemiluminescence in an automated analyzer.
Force-velocity relationship of shoulder muscles pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Force-velocity relationship of shoulder muscles will be assessed by a linear encoder.
Force-velocity relationship of shoulder muscles post-supplementation | Within 2 weeks after the end of supplementation.
  Force-velocity relationship of shoulder muscles will be assessed by a linear encoder.
Maximal grip strength pre-supplementation | Within 2 weeks before the beginning of supplementation
  Maximal grip strength will be assessed by a hand dynamometer
Maximal grip strength post-supplementation | Within 2 weeks after the end of supplementation.
  Maximal grip strength will be assessed by a hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Mougios, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Laboratory of Evaluation of Human Biological Performance, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No